CLINICAL TRIAL: NCT04500951
Title: Evaluation and Improvement of Rest Activity Cycles and Rest Quality in Patients With Severe Acquired Brain Injury
Brief Title: OPTImized RESTing Environments in Rehabilitation
Acronym: OPTIREST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Descriptive studies were published based on this record. Randomized Controlled time-series study was discontinued due to infeasability. Descriptive time-series studies and methodological studies have been published.
Sponsor: University of Aarhus (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Simon Svanborg Kjeldsen, PhD Student, University of Aarhus
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 80; 1-10-72-32-18 (Other: Regional Ethics comitee); 1-10-72-32-18 (Other: Data protection agency)
Record Dates: First submitted 2020-05-05; First posted 2020-08-06 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Acquired Brain Injury
Keywords: Quality of rest; Daytime resting periods; Accelerometry; Electrocardiography
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Intervention Model Description: A Randomized controlled time-series study. A Randomized controlled time-series study. Randomization to either SR or ORE for each of the 9 resting periods during a three-day recording session. A period of three days will allow collection of sufficient data. This will also allow the analysis to take the random effects of time and weekday into account.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimized resting environment (Experimental): The optimized resting environment will consist of the following complex intervention.
  * Technically assisted noise control in regards of alarms in the patient room
  * Visual signing reminding staff that the patient is not to be disturbed during rest
  * Individual optimization of room environment according to information received from relatives
  * Individual optimization of room environment and positioning according to systematized knowledge on best practice in the intervention ward including auditory and visual stimuli
  Interventions: Other: Optimized resting environment
- Standard resting environment (Other): Standard resting environment, will consist of a basic positioning either reclined in bed or reclined in wheelchair according to regular procedures of the ward.
  Interventions: Other: Standard resting environment

INTERVENTIONS:
Other: Optimized resting environment — Alarms from feeding pumps will be relayed to the nurse call system for all intervention periods. Alternatively meals will be timewise reorganized to not interfer with the intervention resting periods. Signs reminding staff not to disturb will be posted for all intervention periods.
  For each patient the close team of rehabilitation professionals will agree upon a guideline suggesting the optimal resting environment for the specific patient. The guideline wil be based on knowledge gathered from relatives on pre-injury preferences. Furthermore, the guideline will be developed based on a toolbox of possible intervention representing best practice. The toolbox has been designed according to the categories of the International Classification of Functioning.
  The intervention will designed individually for each patient.
  Arms: Optimized resting environment
Other: Standard resting environment — The control condition, standard resting environment, will consist of a basic positioning either reclined in bed or reclined in wheelchair according to regular procedures of the ward. Pressure ulcers and positioning believed to induce pain will be avoided.
  Arms: Standard resting environment

SUMMARY:
This study investigates whether an individually designed environment can support and improve the quality of daytime resting periods in in-hospital neurorehabilitation of patients suffering severe acquired brain injury.

The effect of a individually optimized resting environment will be tested against a standard resting environment.

DETAILED DESCRIPTION:
Aim:

The aim is to identify differences in quality of rest as reflected by clinical evaluation, pulse rate, motor activity and autonomic balance between the optimized resting environment (ORE) and the standard resting environment (SR).

Method: A Randomized controlled time-series study. Randomization to either SR or ORE for each of the 9 resting periods during a three-day recording session. A period of three days will allow collection of sufficient data. This will also allow the analysis to take the random effects of time and weekday into account. Outcome measures will be differences in mean heart rate during daytime resting periods, aggregated measures of heart rate variability and proportion of resting minutes according to accelerometry.

ELIGIBILITY:
Inclusion Criteria:

* Severe Acquired brain injury
* >= 18 years
* Relatives/Surrogate can give informed consent
* Classified as being ≤ 7 on the level of cognitive functions scale (also known as Rancho Los Amigos Scale)

Exclusion Criteria:

* Admitted due to polyneuropathies e.g. Guillain-Barré
* Terminal illness
* Spinal lesions
* Expected stay < 3 weeks
* Paroxysmal Sympathetic Hyperactivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation of quality of rest | Measurement represent the evaluated quality of rest for the duration of the resting period. Duration of resting periods will be varying according to the needs of the patients for each resting period. Estimated to be 30 minutes to 2½ hours.
  A five option categorical scale going from "really bad"-"bad"-"good"-"really good "+ the option of "insufficient information for evaluation". Evaluation is performed by the patient responsible clinician at the end of each resting period. Duration of resting periods will be varying according to the needs of the patients for each resting period.
Actigraphic evaluation of motor rest ratio (MRR) | Continuous data will be aggregated from the duration of each resting period. Duration of resting periods will be varying according to the needs of the patients for each resting period. Estimated to be 30 minutes to 2½ hours.
  Actigraphy will be measured during all resting periods. Epochs of 1 minute will be defined as active or inactive based on previous used limits.
  Motor rest ratio (MRR) defined as the proportions of minutes defined as resting out of all minutes recorded in each resting periods will be used to describe degree of motor rest
Heart rate variability: LF band of the power spectrum of a 256 hz ECG recording | Continuous data will be aggregated from the duration of each resting period. Duration of resting periods will be varying according to the needs of the patients for each resting period. Estimated to be 30 minutes to 2½ hours.
  The mean or median (Depending on distribution) low frequency power spectrum of all epochs for the duration of the resting periods will be used to characterize the balance in the autonomous nervous system.
Heart rate variability: HF band of the power spectrum of a 256 hz ECG recording | Continuous data will be aggregated from the duration of each resting period. Duration of resting periods will be varying according to the needs of the patients for each resting period. Estimated to be 30 minutes to 2½ hours.
  The mean or median (Depending on distribution) High frequency power spectrum of all epochs for the duration of the resting periods will be used to characterize the balance in the autonomous nervous system.
Heart rate variability: LF/HF ratio of the power spectrum of a 256 hz ECG recording | Continuous data will be aggregated from the duration of each resting period. Duration of resting periods will be varying according to the needs of the patients for each resting period. Estimated to be 30 minutes to 2½ hours.
  The mean or median (Depending on distribution) LF/HF ratio of all epochs for the duration of the resting periods will be used to characterize the balance in the autonomous nervous system.
Heart rate variability: SDNN a time domain estimate of heart rate variability from of a 256 hz ECG recording | Continuous data will be aggregated from the duration of each resting period. Duration of resting periods will be varying according to the needs of the patients for each resting period. Estimated to be 30 minutes to 2½ hours.
  The mean or median (Depending on distribution) SDNN of all epochs for the duration of the resting periods will be used to characterize the balance in the autonomous nervous system.
Heart rate | Continuous data will be aggregated from the duration of each resting period. Duration of resting periods will be varying according to the needs of the patients for each resting period. Estimated to be 30 minutes to 2½ hours.
  The mean/median heart rate of a 0.2 hz reported heart rate as measured by the monitor system Mindray nseries TM80.
Respiratory rate | Continuous data will be aggregated from the duration of each resting period. Duration of resting periods will be varying according to the needs of the patients for each resting period. Estimated to be 30 minutes to 2½ hours.
  The mean/median respiratory rate of a 0.2 hz reported respiratory rate as extrapolated by the monitor system Mindray nseries TM80 from a 256 hz ecg.

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen F Nielsen, MD DMSc, Study Director — Hammel Neurorehabilitation Centre and University Research Clinic
Locations (1):
- Regionshospitalet Hammel Neurocenter, Hammel, Denmark

IPD SHARING:
Plan to Share IPD: No
Not possible due to GDPR and ethics considerations

REFERENCES:
- See also: Aarhus University project description site — https://pure.au.dk/portal/da/projects/evaluation-and-improvement-of-rest-activity-cycles-and-quality-of-rest-in-patients-with-severe-acquired-brain-injury(a4948657-bc8b-455b-bfeb-189e19bf0af3).html